CLINICAL TRIAL: NCT07380282
Title: Additional Effects of Strength Training With Otago Exercises on Actual and Perceived Balance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/17
Record Dates: First submitted 2025-12-29; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Aged; Postural Balance; Exercise Therapy; Muscle Strength; Resistance Training; Fall Prevention
Keywords: Older adults; Falls prevention; Otago Exercise Program; Strength training; Balance confidence; Postural stability; actual balance; perceived balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago with strengthening exercise (Experimental): The Otago Exercise Program (OEP) is an evidence-based fall-prevention program designed for older adults, focusing on improving strength, balance, and mobility. It emphasizes lower-limb strengthening of key muscle groups such as the quadriceps, hamstrings, hip abductors, and ankle muscles through exercises like seated leg extensions, heel raises, sit-to-stand, and standing leg curls. The balance component includes static and dynamic activities such as tandem walking, single-leg stance, sideways walking, backward walking, and stair stepping, with gradual progression to safely challenge postural control. In this study, strengthening exercises are integrated with the OEP to enhance overall effectiveness. The program is delivered three times per week, with each session lasting 40-45 minutes over an 8-week period. This combined intervention aims to improve balance, reduce fall risk, and increase confidence during daily functional activities among older adults.
  Interventions: Procedure: Otago Exercise with Strengthening exercise
- Otago (Other): Otago exercise plan is comprisedset of 14 exercises including strengthening and balance exercises. The strenghtening exercises include strengthening of Knee Flexors, Knee Extensors, Hip-abductors Ankle dorsiflexors and ankle planter flexors and the balance exercises include following activities: Knee Bends Backward Walking, Walking and Turning Around, Sideways Walking, Tandem Stance, Tandem Walk, One Leg stance, Heel Walking, Toe Walking, Heel toe walk backwards, Sit to stand, Stair Walking These exercises will be performed for a duration 6 weeks and will be performed thrice for a period of 40/50 minutes
  Interventions: Procedure: Otago Exercise Program

INTERVENTIONS:
Procedure: Otago Exercise with Strengthening exercise — The experimental group participated in an 8-week training program, conducted three times per week with 30-45-minute sessions. Each session began with a 5-10 minute warm-up, including dynamic stretching, marching in place, and joint mobility exercises. The program included progressive strength and balance training, starting with light or no resistance and gradually increasing to moderate-high intensity (45-75% of 1RM). Exercises included seated leg extensions, standing leg curls, sit-to-stand, heel raises, step-ups, wall push-ups, and functional movements such as sideways walking, backward walking, and obstacle walking. Balance training involved static and dynamic tasks, including tandem stance, single-leg stance, functional reach, and dynamic walking with turns. Exercise intensity and complexity progressed throughout the program while maintaining safe rest intervals. Each session concluded with a 5-10 minute cool-down, consisting of lower-limb stretching (quadriceps, hamstrings, calves
  Arms: Otago with strengthening exercise
Procedure: Otago Exercise Program — The training program was conducted three times a week, with 30-45-minute sessions. Each session began with a 5-7 minute warm-up (marching in place, ankle circles, shoulder rolls). During Weeks 1-2, participants performed sit-to-stand, heel raises, and seated knee extensions (2 × 10), along with sideways walking (5 m, 2-3 reps) and static balance progressing from feet together to tandem stance. In Weeks 3-4, difficulty increased with sit-to-stand (3 × 10), heel-to-toe walking (5 m), backward walking (3-5 m), single-leg stance (10-15 s), and step-ups (2 × 10). During Weeks 5-6, exercises included wall push-ups, heel raises on a step, dynamic walking with 180° turns, functional reach, and eyes-closed balance tasks. In Weeks 7-8, advanced balance tasks were added, including weighted sit-to-stand, single-leg stance with arm movements, obstacle walking, higher step-ups, and dynamic tandem walking. Each session ended with a 5-7 minute cool-down of lower-limb stretching and breathing exercises
  Arms: Otago

SUMMARY:
This study, titled "Additional Effects of Strength Training with Otago Exercises on Actual and Perceived Balance in Older Adults", explores strategies to reduce fall risks in the elderly. Falls are a major health concern, often causing injuries, loss of mobility, and reduced quality of life. The Otago Exercise Program (OEP) has been proven effective in improving lower-limb strength and balance, but it primarily focuses on these areas without addressing overall muscle strengthening.

The research aims to assess whether integrating additional strength training with OEP can enhance both actual balance (measured through static and dynamic stability tests) and perceived balance (confidence in avoiding falls). Using a randomized controlled trial, 34 participants aged 60 and above will be recruited and divided into two groups: one receiving OEP alone, and the other combining OEP with structured strength training. Tools such as the Berg Balance Scale, Functional Reach Test, Fall Efficacy Scale, and CONFbal Scale will measure outcomes.

The intervention will last eight weeks, with progressive resistance and balance tasks. Findings are expected to demonstrate improved mobility, reduced fear of falling, and greater confidence among participants receiving combined training. This research addresses a significant gap in geriatric rehabilitation and aims to inform cost-effective, evidence-based strategies for fall prevention, ultimately enhancing independence and quality of life in older adults.

DETAILED DESCRIPTION:
Falls among older adults represent a critical public health issue, often resulting in injuries, loss of independence, and reduced quality of life. Globally, up to 35% of people over 65 experience falls annually, with risk increasing as age advances. The major contributors are muscle weakness and impaired balance, often linked to sarcopenia, an age-related decline in muscle mass and strength. These deficits compromise postural stability, mobility, and coordination, increasing vulnerability to recurrent falls and associated complications.

The Otago Exercise Program (OEP) is a recognized intervention for fall prevention, focusing on lower-limb strengthening and balance training. Evidence shows it reduces fall rates significantly, yet its scope remains limited to balance and limb strength, overlooking broader muscular demands. Integrating structured strength training with OEP may enhance outcomes by improving static and dynamic stability, muscle power, and confidence in daily tasks. Addressing both physical and psychological factors, such an approach can reduce fall-related injuries, foster independence, and improve quality of life in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 60 years and above.
* Mini-Mental State Examination (MMSE) score of 24 or higher (sufficient cognitive ability to participate).
* Individuals able to ambulate independently or with minimal assistance (e.g., cane).
* Those who have not participated in a structured balance or strengthening program in the past 3 months.
* Participants able to provide informed consent and adhere to the intervention protocol.

Exclusion Criteria:

* Severe musculoskeletal or neurological conditions limiting mobility (e.g., advanced arthritis, stroke with significant residual deficits).
* Sensory disabilities affecting vision, hearing, or vestibular function.
* Structural defects in extremities.
* Fracture in the past year.
* Unstable systemic pathology, recent surgery, or cancer diagnosis/treatment within the past 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Actual Balance | 8 weeks
  The 1st primary outcome is the improvement in actual balance Berg Balance Scale (BBS) Score range: 0-56
  Cut-off values:
  * 41-56 Low fall risk
  * 21-40 Medium fall risk
  * 0-20 High fall risk < 45 = Increased risk of falls
Functional Reach | 8 Weeks
  Functional Reach Test Measured in centimeters (cm)
  Cut-off values:
  * > 25 cm Low fall risk
  * 15-25 cm Moderate fall risk
  * < 15 cm High fall risk < 18.5 cm = Increased fall risk in older adults

SECONDARY OUTCOMES:
Perceived balance | 8 weeks
  : Falls Efficacy Scale - International (FES-I) Score range: 16-64
  Cut-off values:
  * 16-19 Low concern about falling
  * 20-27 Moderate concern
  * 28-64 High concern / high fall risk
Perceived Balance | 8 weeks
  CONFbal scale
  Cut-off value:
  * < 67% → High risk of falling
  * ≥ 67% → Low risk of falling Widely used for community-dwelling older adults

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan